CLINICAL TRIAL: NCT02977481
Title: Ear Temperature, Measured With 3. Generation Tympanic Thermometers as Predictor of Rectal Temperature in the Emergency Department Population
Brief Title: Ear Temperature as Predictor of Rectal Temperature Measured With Modern Devices in the Emergency Department.
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christian Backer Mogensen, asst professor, University of Southern Denmark
Other Study IDs: SHS-ED-11-2016
Record Dates: First submitted 2016-11-18; First posted 2016-11-30 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Fever
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Ear thermometers are often requested to be used rather than rectal thermometer (gold standard) for measuring the body temperature, as this method is faster and more user friendly. Former ear thermometers did not meet the required standards of accuracy for clinical use. However, a new generation of ear thermometers have been developed and widely used in the Emergency departments in Denmark. The devices have only been evaluated in two studies on adult populations, with conflicting results.

This cross-sectional study will examine patients by measuring both ear and rectal temperature in the same patient at the same time on admission to an emergency department, to evaluate if temperature measured in the ear can be used as the standard temperature measurement.

ELIGIBILITY:
Inclusion Criteria:

* admission to emergency department

Exclusion Criteria:

* no rectum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 600 adult patients admitted to emergency department
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The Body Temperature in Celcius degrees | Up to 24 hours after arrival to Emergency Department

CONTACTS AND LOCATIONS:
Locations (1):
- Aabenraa Sygehus Emergency Department, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mogensen CB, Vilhelmsen MB, Jepsen J, Boye LK, Persson MH, Skyum F. Ear measurement of temperature is only useful for screening for fever in an adult emergency department. BMC Emerg Med. 2018 Dec 3;18(1):51. doi: 10.1186/s12873-018-0202-5. PMID 30509206